CLINICAL TRIAL: NCT02325115
Title: Validation of the French Warwick-Edinburgh Mental Well-being Scale (WEMWBS) in Both Non-clinical and Clinical Populations
Brief Title: Validation of the French Warwick-Edinburgh Mental Well-being Scale (WEMWBS)
Status: Completed | Type: Observational
Sponsor: Hôpital le Vinatier (Other)
Collaborators: Institut de Recherche Biomedicale des Armees (Other Government); Fondation de France (Other); Université d'Auvergne (Other); Australian Catholic University (Other)
Responsible Party: Principal Investigator, Nicolas FRANCK, Pr, Professor, Hôpital le Vinatier
Other Study IDs: 2010-A00212-37
Record Dates: First submitted 2014-12-17; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Human Characteristics; Attitude to Health
Keywords: well-being, mental health, schizophrenia, quality of life
MeSH Terms: conditions — Psychological Well-Being; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- students (STUD): The STUD population was a convenient sample of 75 first year students (51 females and 24 males); with 45 from a School of Business Management and 30 from a medical university.
- working adults (WORK): The WORK population was also a convenient sample of 113 (63 females and 256 males) working adults including 217 soldiers from Paris Fire Brigade, 93 nurses and 9 individuals from a research laboratory.
- remitted schizophrenia (PRS): The PRS population was comprised of 121 remitted schizophrenia patients (39 females and 82 males) who were all clients of the rehabilitation centre for psychotic disorders (Le Vinatier hospital),

SUMMARY:
Background: Despite current popularity, positive mental health is under researched. This is possibly due to a lack of consensus on appropriate measuresThe Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) is a 14 positively phrased Likert-style list of items developed to measure mental well-being. Its validation has been internationally explored. This report presents the French validation of the WEMWBS (F-WEMWBS) in non-clinical and clinical populations.

Methods: Two non-clinical populations comprised of 319 working adults (WORK), and 75 students (STUD), and one clinical population of 121 patients with remitted schizophrenia (PRS) were included in the validation study. Participants completed the F-WEMWBS as well as complementary measures of psychological constructs potentially related to well-being.

DETAILED DESCRIPTION:
Three different populations participated in the study: two non-clinical populations composed of students (STUD), and working adults (WORK) and one clinical population comprised of patients with remitted schizophrenia (PRS). The STUD population was a convenient sample of 75 first year students (51 females and 24 males); with 45 from a School of Business Management and 30 from a medical university. The WORK population was also a convenient sample of 113 (63 females and 256 males) working adults including 217 soldiers from Paris Fire Brigade, 93 nurses and 9 individuals from a research laboratory. The PRS population was comprised of 121 remitted schizophrenia patients (39 females and 82 males) who were all clients of the rehabilitation centre for psychotic disorders (Le Vinatier hospital), situated in Lyon, France.

ELIGIBILITY:
Inclusion Criteria:

* For STUD and WORK, there were two criteria to be included in the study: (i) , not undergoing medical treatment for psychological issues at the time of the study and (ii) and not having been part of a stress management program prior to recruitment for the current study.
* For PRS, there were three criteria to be included in the study: (i) a DSM-IVR diagnosis of schizophrenia as confirmed by the Mini International Neuropsychiatric Interview for DSM-IV (MINI; 14); (ii) age between 18 and 65 years; and (iii) being clinically stable (i.e. not having required hospitalization or increases in medication as a result of an exacerbation of acute symptoms over the previous three months).

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three different populations participated in the study: two non-clinical populations composed of students (STUD), and working adults (WORK) and one clinical population comprised of patients with remitted schizophrenia (PRS).
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) | Baseline and 2 months